CLINICAL TRIAL: NCT01013532
Title: A Multicenter, Double Blind, Factorial Design, Phase IV Trial to Compare the Efficacy and Safety of Cilostazol Long-term Treatment With Aspirin in Ischemic Stroke Patients With High Risk of Cerebral Hemorrhage for the Prevention of Cerebral Hemorrhage and Cardiovascular Events and to Compare the Preventive Effect of Probucol in the Same Patient Group With Non-drug User Group for the Prevention of Cardiovascular Events
Brief Title: PreventIon of CArdiovascular Events in iSchemic Stroke Patients With High Risk of Cerebral HemOrrhage
Acronym: PICASSO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sun U. Kwon, Professor, Asan Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PICASSO
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Brain Ischemia; Intracranial Hemorrhages
Keywords: Ischemic Stroke; Intracranial Hemorrhage; Cilostazol; Probucol
MeSH Terms: conditions — Brain Ischemia; Intracranial Hemorrhages; Ischemic Stroke | interventions — Cilostazol; Probucol; Aspirin; Ankle Brachial Index

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cilostazol+ Probucol (Experimental): 100mg cilostazol bid plus probucol plus placebo of aspirin
  Interventions: Drug: Cilostazol; Drug: Probucol; Drug: placebo of aspirin; Device: ankle-brachial index (ABI); Device: intima-medial thickness (IMT); Device: new asymptomatic brain hemorrhage; Device: new ischemic lesions on follow-up FLAIR images
- Aspirin + Probucol (Active Comparator): aspirin plus placebo cilostazol plus probucol
  Interventions: Drug: Probucol; Drug: Aspirin; Drug: placebo of cilostazol; Device: ankle-brachial index (ABI); Device: intima-medial thickness (IMT); Device: new asymptomatic brain hemorrhage; Device: new ischemic lesions on follow-up FLAIR images
- Cilostazol (Experimental): cilostazol plus placebo of aspirin
  Interventions: Drug: Cilostazol; Drug: placebo of aspirin; Device: ankle-brachial index (ABI); Device: intima-medial thickness (IMT); Device: new asymptomatic brain hemorrhage; Device: new ischemic lesions on follow-up FLAIR images
- Aspirin (Active Comparator): aspirin plus placebo of cilostazol
  Interventions: Drug: Aspirin; Drug: placebo of cilostazol; Device: ankle-brachial index (ABI); Device: intima-medial thickness (IMT); Device: new asymptomatic brain hemorrhage; Device: new ischemic lesions on follow-up FLAIR images

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100mg bid
  Other Names: Pletaal produced by Korea Otsuka Pharmaceutical company
  Arms: Cilostazol; Cilostazol+ Probucol
Drug: Probucol — Probucol 250mg bid
  Other Names: Probucol is produced by Otsuka Pharmaceutical
  Arms: Aspirin + Probucol; Cilostazol+ Probucol
Drug: Aspirin — Aspirin 100mg qd
  Arms: Aspirin; Aspirin + Probucol
Drug: placebo of cilostazol — same shape and size of active cilostazol
  Arms: Aspirin; Aspirin + Probucol
Drug: placebo of aspirin — same size and shape of active aspirin 100mg
  Arms: Cilostazol; Cilostazol+ Probucol
Device: ankle-brachial index (ABI) — measurement of ABI every years during follow up
Device: intima-medial thickness (IMT) — ultrasound measured IMT of both common carotid arteries
  Other Names: change of maximal IMT and mean IMT
Device: new asymptomatic brain hemorrhage — asymptomatic macrobleedings or microbleedings on GRE images
Device: new ischemic lesions on follow-up FLAIR images — any new ischemic lesions

SUMMARY:
Through this study, the investigators are to prove that Cilostazol effectively prevent cardiovascular events in ischemic stroke patients with high risk of cerebral hemorrhage, along with no significant increase in the risk of occurrence of hemorrhagic side effects.

The primary hypothesis of this study is; Cilostazol alone or with probucol will reduce the risk of cerebral hemorrhage without increase of cardiovascular events compared to aspirin in the ischemic stroke patients with symptomatic or asymptomatic old cerebral hemorrhage.

This study will prove the superiority of cilostazol on the prevention of cerebral hemorrhagic events without increasing the cardiovascular events against aspirin and the superiority of probucol on the prevention of overall cardiovascular events.

DETAILED DESCRIPTION:
It has been generally accepted that 'old age' and 'hypertension' may be risk factors not only for cerebral infarction but also for cerebral hemorrhage. Usually 40 to 60 percent of recurrent strokes after cerebral hemorrhage cases are cerebral infarction; and 5 to 10 percent of recurrent stroke after cerebral infarction cases are cerebral hemorrhage.

Consequently, for the reasons described above, hemorrhagic side effects including cerebral hemorrhage have been a great concern, in the usage of antiplatelet agent or anticoagulant for the secondary prevention in the patients with cerebral infarction.

It is reported that the occurrence of cerebral hemorrhage tends to increase in cases of accompanying lacunar infarction which occurs more frequently in Asians than in Westerners, or periventricular ischemic change which increasingly occurs with ageing. Accordingly, the point is that the occurrence of cerebral hemorrhage should be primarily considered in the treatment of cerebral infarction, along with the phenomenon of an ageing population both in Asian countries including Korea.

Nevertheless, so far there has been no clinical research regarding secondary prevention of stroke, particularly considering the risk of occurrence of hemorrhage in cerebral infarction cases. However, according to a recent study, when phosphodiesterase inhibitors including Cilostazol are used independently, or in combination with aspirin, secondary prevention can be improved without increasing the occurrence of hemorrhagic side effects.

Considering this, if it is proved that the agent, Cilostazol, could decrease the risk of occurrence of stoke, along with no significant increase in the risk of occurrence of hemorrhagic side effects, by selecting a patent group with a high risk of cerebral hemorrhage, the agent (Cilostazol) may be recognized as an unique antiplatelet agent applicable to old-aged patient with cerebral infarction who have a certain risk of cerebral hemorrhage.

* High risk of cerebral hemorrhage is defined as presence of history of cerebral hemorrhage with appropriate neuroimage findings or presence of asymptomatic old cerebral hemorrhage findings(equal or more than 8mm) or multiple microbleeds on the GRE images.
* 1600 ischemic stroke patients with high risk of cerebral hemorrhage will be recruited and they are randomized into four groups (cilostazol plus probucol, aspirin plus probucol, cilostazol and aspirin) by 2X2 factorial design.
* IMT and ABI will be measured every year during follow-up period and the results will be compared with the baseline data. The change of IMT and ABI will be analyzed with the occurrence of cardiovascular events.
* The study will finish at least 1 year after the recruit of 1600th patients. Until the finish, all patients will continuously take study medications and visit every 3months at the study site.
* Brain MRI including FLAIR and GRE will be done at the final visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transient ischemic attack (TIA) or ischemic stroke within 180 days prior to screening - Adult aged 20 years or older
* High risk of hemorrhagic stroke (history of intracranial hemorrhage or imaging evidence of previous intracranial hemorrhage)
* Informed consent

Exclusion Criteria:

* Clinical diagnosis of myocardial infarction or coronary intervention within 4 weeks
* Bleeding tendency
* Pregnant or breast-feeding woman
* Hemorrhagic stroke within 6 months
* Patient who was taking antithrombotic medication other than aspirin and does not agree to change the previous medication
* Severe cardiovascular disease such as cardiomyopathy or congestive heart failure
* Life expectancy less than one year
* Contraindication to long term aspirin use
* Enrolled in other clinical trial within 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2009-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of cerebral hemorrhage | time since randomization; follow-up period is 1.0 to 5.5 years
Time to the first occurence of composite cardiovascular events | time since randomization; follow-up period is 1.0 to 5.5 years

SECONDARY OUTCOMES:
Time to the first occurrence of stroke | time since randomization; follow-up period is 1.0 to 5.5 years
Time to the first occurrence of ischemic stroke | time since randomization; follow-up period is 1.0 to 5.5 years
Time to the first occurence of myocardial infarction | time since randomization; follow-up period is 1.0 to 5.5 years
Time to the first occurence of other designated vascular events | time since randomization; follow-up period is 1.0 to 5.5 years

OTHER OUTCOMES:
Incidence rate of major and non-major hemorrhagic event | time since randomization; follow-up period is 1.0 to 5.5 years
Rate of asymptomatic hemorrhage in GRE (microhemorrhage or macrohemorrhage) | at final visit, follow-up MRI will be checked at the final visit
Rate of new asymptomatic cerebral infarction lesion in FLAIR | at final visit, follow-up MRI will be checked at the final visit
Change of ankle-brachial index | at final visit;follow-up period is 1.0 to 5.5 years
The effect of the size of common carotid artery(CCA) including plaque on the occurrence of cardiovascular events | at final visit;follow-up period is 1.0 to 5.5 years
Time to all deaths including vascular and non-vascular deaths | time since randomization; follow-up period is 1.0 to 5.5 years
Incidence rate of dementia diagnosed after initiation of the trial | time since randomization; follow-up period is 1.0 to 5.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sun U. Kwon, MD, PhD, Principal Investigator — Departement of Neurology, Asan Medical Center
Locations (71):
- China (4):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong, Hong Kong
  - United Christian Hospital, Hong Kong, Hong Kong
  - Prince of Wales Hospital, Shatin, NT, Hong Kong
- Philippines (4):
  - Manila Doctors Hospital, Manila
  - University of Santo Tomas, Manila
  - The Medical City, Pasig
  - St. Luke's Medical Center, Quezon City
- South Korea (63):
  - Wallace Memorial Baptist Hospital, Busan, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan, Chungcheongnam-do
  - Keimyung University Dongsan Center, Daegu, Daegu
  - Daegu Fatima Hospital, Daegu, Daegu
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Kwandong University College of Medicine Myongji Hospital, Gyeonggi-do, Goyang
  - Gyeongsang National University Hospital, Jinju, Gyengsangnam-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - National Health Insurance Corporation Ilsan Hoapital, Goyang-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - Samsung changwon Medical Center, Changwon, Gyeongsangnam-do
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chang Won Fatima hospital, Changwon, Kyeongsangnam-do
  - Dongguk University International Hospital, Goyang, Kyoungki-do
  - Hallym University Sacred Heart Hospital, Anyang, Kyunggi
  - Seoul National University Bundang Hospital, Seongnam, Kyunggi
  - Ajou University Hospital, Suwon, Kyunggi
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Kosin University Gospel Hospital, Busan
  - Inje University Pusan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Dong-A University Hospital, Busan
  - Eulji University Hospital, Daejeon
  - Dongsan Medical Center, Deagu
  - Kyungpook National University Hospital, Deagu
  - Yeungnam University Medical Center, Deagu
  - Deagu Catholic University Hospital, Deagu
  - Chungnam National University Hospital, Deajeon
  - Deajeon St.Mary's Hospital, The Catholic University of Korea, Deajeon
  - Chosun University Hospital, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hoapital, Incheon
  - Inha University Hospital, Inchon
  - National Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Hanyang University Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Hallym University, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul St.Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Konkuk Univ. Hospital, Seoul
  - St. Mary's Hospital, Seoul
  - Hangang Sacred Heart Hospital, Seoul
  - Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Borame Hospital, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Eulji Hospital, Seoul
  - Chung-Ang University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Park JH, Lee J, Kwon SU, Sung Kwon H, Hwan Lee M, Kang DW. Elevated Pulse Pressure and Recurrent Hemorrhagic Stroke Risk in Stroke With Cerebral Microbleeds or Intracerebral Hemorrhage. J Am Heart Assoc. 2022 Feb;11(3):e022317. doi: 10.1161/JAHA.121.022317. Epub 2021 Nov 15. PMID 34779245
- [Derived] Cho KH, Kwon SU, Lee JS, Yu S, Cho AH. Newly diagnosed diabetes has high risk for cardiovascular outcome in ischemic stroke patients. Sci Rep. 2021 Jun 21;11(1):12929. doi: 10.1038/s41598-021-92349-y. PMID 34155277
- [Derived] Park HK, Lee JS, Kim BJ, Park JH, Kim YJ, Yu S, Hwang YH, Rha JH, Heo SH, Ahn SH, Seo WK, Park JM, Lee JH, Kwon JH, Sohn SI, Jung JM, Kwon SU, Hong KS; PICASSO investigators. Cilostazol versus aspirin in ischemic stroke with cerebral microbleeds versus prior intracerebral hemorrhage. Int J Stroke. 2021 Dec;16(9):1019-1030. doi: 10.1177/1747493020941273. Epub 2020 Jul 14. PMID 32664827
- [Derived] Lee EJ, Kwon SU, Park JH, Kim YJ, Hong KS, Yu S, Hwang YH, Lee JS, Lee J, Rha JH, Heo SH, Ahn SH, Seo WK, Park JM, Lee JH, Kwon JH, Sohn SI, Jung JM, Kim HY, Kim EG, Kim SH, Cha JK, Park MS, Nam HS, Kang DW; PICASSO Investigators. Changes in High-Density Lipoprotein Cholesterol and Risks of Cardiovascular Events: A Post Hoc Analysis from the PICASSO Trial. J Stroke. 2020 Jan;22(1):108-118. doi: 10.5853/jos.2019.02551. Epub 2020 Jan 31. PMID 32027796
- [Derived] Kim BJ, Kwon SU, Park JH, Kim YJ, Hong KS, Wong LKS, Yu S, Hwang YH, Lee JS, Lee J, Rha JH, Heo SH, Ahn SH, Seo WK, Park JM, Lee JH, Kwon JH, Sohn SI, Jung JM, Navarro JC, Kim HY, Kim EG, Kim S, Cha JK, Park MS, Nam HS, Kang DW; PICASSO Investigators. Cilostazol Versus Aspirin in Ischemic Stroke Patients With High-Risk Cerebral Hemorrhage: Subgroup Analysis of the PICASSO Trial. Stroke. 2020 Mar;51(3):931-937. doi: 10.1161/STROKEAHA.119.023855. Epub 2019 Dec 20. PMID 31856691
- [Derived] Kim BJ, Lee EJ, Kwon SU, Park JH, Kim YJ, Hong KS, Wong LKS, Yu S, Hwang YH, Lee JS, Lee J, Rha JH, Heo SH, Ahn SH, Seo WK, Park JM, Lee JH, Kwon JH, Sohn SI, Jung JM, Navarro JC, Kang DW; PICASSO investigators. Prevention of cardiovascular events in Asian patients with ischaemic stroke at high risk of cerebral haemorrhage (PICASSO): a multicentre, randomised controlled trial. Lancet Neurol. 2018 Jun;17(6):509-518. doi: 10.1016/S1474-4422(18)30128-5. PMID 29778364
- [Derived] Park TH, Lee JS, Park SS, Ko Y, Lee SJ, Lee KB, Lee J, Kang K, Park JM, Choi JC, Kim DE, Cho YJ, Kim JT, Kim DH, Cha JK, Han MK, Lee J, Oh MS, Yu KH, Lee BC, Bae HJ, Hong KS. Safety and efficacy of intravenous recombinant tissue plasminogen activator administered in the 3- to 4.5-hour window in Korea. J Stroke Cerebrovasc Dis. 2014 Aug;23(7):1805-12. doi: 10.1016/j.jstrokecerebrovasdis.2014.04.027. Epub 2014 Jun 21. PMID 24957314